CLINICAL TRIAL: NCT05014360
Title: A Phase 1b Study to Evaluate the Efficacy and Safety of JNJ-64251330, a Janus Kinase (JAK) Inhibitor, in Participants With Familial Adenomatous Polyposis
Brief Title: A Study of JNJ-64251330 in Participants With Familial Adenomatous Polyposis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR109012; 2021-001068-16 (EudraCT Number); 64251330COR1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-08-13; First posted 2021-08-20 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-06

CONDITIONS: Adenomatous Polyposis Coli
MeSH Terms: conditions — Adenomatous Polyposis Coli

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- JNJ-64251330 (Experimental): Participants will receive oral dose of JNJ-64251330 twice daily for 24 Weeks.
  Interventions: Drug: JNJ-64251330

INTERVENTIONS:
Drug: JNJ-64251330 — JNJ-64251330 tablets will be administered orally.
  Other Names: Lorpucitinib

SUMMARY:
The purpose of this study is to determine the effect of JNJ-64251330 in participants with Familial Adenomatous Polyposis (FAP) on colorectal polyp burden (sum of the polyp diameters).

DETAILED DESCRIPTION:
Familial adenomatous polyposis (FAP) is the most common polyposis syndrome. It is an autosomal dominant inherited disorder characterized by the early onset of hundreds to thousands of adenomatous polyps throughout the colon. JNJ-64251330 (lorpucitinib) is an oral, small molecule, potent pan-janus kinase (JAK) inhibitor that blocks phosphorylation of Signal Transducer and Activator of Transcription (STAT) proteins. pSTAT induces transcription of multiple genes involved in the progression of inflammatory disease. JNJ-64251330 has chemical properties that limits the amount of drug in the blood while delivering the drug to the tissues of the gut. Local inhibition of JAK in the gut may present a promising method to treat inflammatory diseases of the intestinal tract, such as FAP. The study consists of 3 phases: screening phase (30 days) a treatment phase (24 weeks), and follow-up visit (up to 30 days after last dose of study drug). The total duration of the study will be up to 32 weeks. Study evaluations will include efficacy via endoscopies, safety (monitoring of adverse events (AE), serious adverse events (SAEs), events of infections including tuberculosis (TB), clinical laboratory blood tests (complete blood count and serum chemistries), vital signs, and concomitant medication review), pharmacokinetics, pharmacodynamic and biomarkers evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Genetic diagnosis of classical familial adenomatous polyposis (FAP) (adenomatous polyposis coli [APC] germline mutation or obligate carrier) with disease involvement of the colorectum
* At least 6 polyps greater than or equal to (>=) 2 millimeters (mm) in diameter in the rectum or colon
* A female participant of childbearing potential must have a negative highly sensitive pregnancy test at screening and within 72 hours prior to the first dose of study drug and must agree to further pregnancy tests during the study
* A male participant must agree not to donate sperm for the purpose of reproduction during the study and for a minimum of 90 days after receiving the last dose of study drug
* Must sign an informed consent form (ICF) indicating he or she understands the purpose of the study and procedures required for the study and is willing to participate in the study. Consent is to be obtained prior to the initiation of any study-related tests or procedures that are not part of standard of care for the participant's disease

Exclusion Criteria:

* Use of non-steroidal anti-inflammatory drugs (example, aspirin, ibuprofen) exceeding 5 days per month or exceeding the nonprescription dose, unless the participant completes a 4-week washout period prior to the first dose of study drug
* Treatment with other FAP-directed drug therapy (including sulindac or celecoxib), unless completes a 4-week washout period prior to the first dose of study drug
* History of human immunodeficiency virus (HIV)
* History of severe, progressive, or uncontrolled renal, genitourinary, hepatic, hematologic, endocrine, cardiac, vascular, pulmonary, rheumatologic, neurologic, psychiatric, or metabolic disturbances, or signs and symptoms thereof
* A history of, or ongoing, chronic or recurrent infectious disease including latent or active tuberculosis (TB)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Percentage Change from Baseline in Colorectal Polyp Burden for all Polyps at Week 24 | Baseline and Week 24
  Percentage change from baseline in colorectal polyp burden for all polyps (the sum of the polyp diameters) at Week 24 will be reported.
Percentage Change from Baseline in Colorectal Polyp Burden for Polyps >=2 mm at Week 24 | Baseline and Week 24
  Percentage change from baseline in colorectal polyp burden (sum of the polyp diameters) for polyps greater than or equal to (>=) 2 millimeters (mm) at Week 24 will be reported.

SECONDARY OUTCOMES:
Percentage Change in Number of Colon Polyps | Baseline and Week 24
  Percentage change in number of colon polyps will be reported.
Percentage Change in Number of Rectal Polyps | Baseline and Week 24
  Percentage change in number of rectal polyps will be reported.
Percentage Change in Number of J-pouch Polyps | Baseline and Week 24
  Percentage change in number of J-pouch polyps (for participants with an ileal pouch-anal anastomosis [IPAA]) will be reported.
Percentage Change in Number of Duodenal Polyps | Baseline and Week 24
  Percentage change in number of duodenal polyps will be reported.
Percentage Change in Colon Polyp Burden for all Polyps, Polyps >=2 mm and Polyps >=5 mm | Baseline and Week 24
  Percentage change in colon polyp burden for all polyps, polyps >=2 mm and polyps >=5 mm will be reported.
Percentage Change in Rectal Polyp Burden for all Polyps, Polyps >=2 mm and Polyps >=5 mm | Baseline and Week 24
  Percentage change in rectal polyp burden for all polyps, polyps >=2 mm and polyps >=5 mm will be reported.
Percentage Change in J-Pouch Polyp Burden for all Polyps, Polyps >=2 mm and Polyps >=5 mm | Baseline and Week 24
  Percentage change in J-Pouch polyp (for participants with an IPAA) burden for all polyps, polyps >=2 mm and polyps >=5 mm will be reported.
Percentage Change in Duodenal Polyp Burden for all Polyps, Polyps >=2 mm and Polyps >=5 mm | Baseline and Week 24
  Percentage change in duodenal polyp burden for all polyps, polyps >=2 mm and polyps >=5 mm will be reported.
Change in International Society for Gastrointestinal Hereditary Tumors (InSiGHT) Polyposis Stage (with and Without Colon) | Baseline and Week 24
  Change in InSiGHT stage will be reported. Various stages are defined as: a) With Colon: Stage 0: 0-10 polyps,all less than [<]5mm); Stage 1: 20-200 polyps,most <5 mm, none, >1 centimeters[cm]; Stage 2: 200-500 polyps,<10 that are >1 cm; Stage 3: 500-1000 polyps or any number if there are 10-50 that are >1 cm and amenable to complete polypectomy; Stage 4: >1000 polyps and/or any polyps grown to confluence and not amenable to simple polypectomy, any invasive cancer; b) Without Colon: Stage 0: 0 -10 polyps, all <5 mm; Stage 1: 10-25 polyps most <5 mm, none >1 cm; Stage 2: 10-25 polyps, any >1 amenable to complete removal; Stage 3: >25 polyps amenable to complete removal, or any incompletely removed sessile polyp, or any evidence of high-grade dysplasia (HGD), even if completely excised; Stage 4: >25 polyps not amenable complete removal, or any incompletely excised sessile polyp showing HGD; any invasive cancer.
Change in Spigelman Stage Score | Baseline and Week 24
  Change in Spigelman stage score will be reported. Spigelman classification system measures risk of developing duodenal cancer in familial adenomatous polyposis (FAP). It has been classified in following stages- Stage 0 (0 points); Stage 1 (1-4 points); Stage 2 (5-6 points); Stage 3 (7-8 points); and Stage 4 (9-12 points). The total score ranges from 0 to 12. The higher the score, the more severe or advanced the FAP disease in the duodenum.
Number of Participants with Adverse Events (AEs) | Up to 32 weeks
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Number of Participants with AEs by Severity | Up to 32 weeks
  Number of participants with AEs by severity will be reported. Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death related to AE.
Plasma Concentration of JNJ-64251330 Over Time | Up to Week 24
  Plasma samples will be analyzed to determine plasma concentrations of JNJ-64251330 using a validated specific, and sensitive liquid chromatography coupled to tandem mass spectrometry detection (LC-MS/MS).
Tissue Concentration of JNJ-64251330 Over Time | Up to Week 24
  Tissue biopsy samples will be analyzed to determine tissue concentrations of JNJ-64251330 using a validated specific, and sensitive LC-MS/MS.
Levels of JAK/STAT Pathway Signaling Effector Proteins including pSTAT-3 Relative to Baseline Levels in Colorectal Polyps | Up to Week 24
  Levels of Pan-janus kinase (JAK)/ signal transducer and activator of transcription (STAT) pathway signaling effector proteins including phosphorylated (p) STAT-3 relative to baseline levels in colorectal polyps will be reported. Polyp and tissue samples will be collected to monitor for changes to the JAK-STAT pathway.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (16):
- United States (5):
  - City of Hope, Duarte, California
  - University of Miami, Miami, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- France (2):
  - Hopital Edouard Herriot - CHU Lyon, Lyon
  - APHM Hopital Timone, Marseille
- Universitatsklinikum Bonn, Bonn, Germany
- Academisch Medisch Centrum Universiteit van Amsterdam, Amsterdam, Netherlands
- Pan American Center for Oncology Trials LLC, Río Piedras, Puerto Rico
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (2):
  - Hosp. Clinic I Provincial de Barcelona, Madrid
  - Clinica Univ. de Navarra, Pamplona

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency